CLINICAL TRIAL: NCT02171637
Title: A Phase I Open Label Dose Escalation Study of Once-daily Oral Treatment With BIBW 2992 for 14 Days in Patients With Advanced Solid Tumors
Brief Title: Dose Escalation Study of Oral Treatment With BIBW 2992 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.1
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Afatinib

ARMS (1):
- BIBW 2992 (Experimental)
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: BIBW 2992 — escalating doses

SUMMARY:
Evaluation of maximum Tolerated Dose (MTD), safety, pharmacokinetics, efficacy of BIBW 2992, pharmacodynamic modulation of biomarkers, correlation of Epidermal Growth Factor Receptor (EGFR) and Human EGF-like Receptor number 2 (HER2) immunohistochemical status with objective tumour responses

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with confirmed diagnosis of advanced, non resectable and / or metastatic solid tumors, of types historically known to express EGFR and/or HER2, who have failed conventional treatment, or for whom no therapy of proven efficacy exists, or who are not amenable to established forms of treatment
* Age 18 years or older
* Life expectancy of at least three (3) months
* Written informed consent given that is consistent with International Conference on Harmonization - Good Clinical Practice (ICH-GCP) guidelines
* Eastern Cooperative Oncology Group (ECOG) performance score 0, 1, or 2
* Patients must have resolution of prior chemo-, hormone, immuno-, or radiotherapy-related toxicities to CTC Grade < 1
* Patients have to be recovered from previous surgery
* Paraffin-embedded tumor material must be accessible for analysis of EGFR and HER2-status.
* The additional 12 patients that were to be recruited at the MTD also had to fulfill the following criterion: Measurable tumor deposits (RECIST: Response Evaluation Criteria in Solid Tumors) by one or more techniques (X-ray, CT, MRI)

Exclusion Criteria:

* Active infectious disease
* Gastrointestinal disorders that might interfere with the absorption of the study drug or chronic diarrhea
* Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol
* Brain metastases requiring therapy as based on clinical symptoms
* Impaired cardiac left ventricular function with resting ejection fraction CTC Grade ≥ 1
* Absolute neutrophil count (ANC) less than 1500 / mm3
* Platelet count less than 100 000 / mm3
* Bilirubin greater than 1.5 mg / dl (> 26 μmol / L, SI unit equivalent)
* Aspartate amino transferase (AST) and / or alanine amino transferase (ALT) greater than three times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal)
* Serum creatinine greater than 1.5 mg / dl (> 132 μmol / L, SI (Systeme International) unit equivalent)
* Women and men who are sexually active and unwilling to use a medically acceptable method of contraception
* Pregnancy or breast-feeding
* Treatment with other investigational drugs; chemotherapy, immunotherapy, radiotherapy or hormone therapy (excluding LHRH agonists, other hormones taken for breast cancer, or bisphosphonates) or participation in another clinical study within the past four weeks before start of therapy or concomitantly with this study
* Patients unable to comply with the protocol
* Active alcohol or drug abuse

RETREATMENT CRITERIA

The patient may be eligible for re-treatment after the previous course finished. The patient will not be eligible if the following criteria are met.

* Patients with clinical signs of disease progression or if an X-ray, CT or MRI was done and the test showed progressive disease
* Cardiac left ventricular function CTC Grade ≥ 2 at any time during the previous course
* Patients fulfilling any of the Exclusion Criteria as mentioned under exclusion criteria on Day 29 of the previous course
* Patients not recovered from any dose-limiting toxicity (DLT) 14 days after the last administration of BIBW 2992 in the previous course. Recovery is defined as a return to baseline level or CTC Grade 1, whichever is higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2003-11; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | up to 28 months
Incidence and intensity of Adverse Events (AE) according to Common Terminology Criteria for Adverse Events (CTCAE) associated with increasing doses of BIBW 2992 | up to 28 months

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) for different time points | up to 384 hours after first drug administration
Predose plasma concentration (Cpre) for different time points | Day 8 and 14
Minimum measured plasma concentration (Cmin) for different time points | up to 384 hours after first drug administration
Maximum measured plasma concentration (Cmax) for different time points | up to 384 hours after first drug administration
Time from dosing to the minimum plasma concentration (tmin) for different time points | up to 384 hours after first drug administration
Time from dosing to the maximum plasma concentration (tmax) for different time points | up to 384 hours after first drug administration
Terminal half-life (t1/2) for different time points | up to 384 hours after first drug administration
Mean residence time after oral administration (MRTpo) for different time points | up to 384 hours after first drug administration
Apparent clearance (CL/F) for different time points | up to 384 hours after first drug administration
Apparent volume of distribution during the terminal phase (Vz/F) for different time points | up to 384 hours after first drug administration
Accumulation ratio (RA) | up to 384 hours after first drug administration
Modulation of biomarker (EGFR, p-EGFR, p-MAPK (mitogen-activated protein kinase), p-Akt, Ki-67, p-27KIP1) in skin biopsies prior to administration of BIBW 2992 and at the end of the first treatment period | Baseline and day 14
Modulation of biomarker (EGFR, p-EGFR, HER2, p-MAPK, p-Akt, Ki-67, p-27KIP1) in tumor biopsies prior to administration of BIBW 2992 and at the end of the first treatment period in 6 or more patients treated at the MTD | Baseline and day 14
Objective tumor responses | every 8 weeks up to 28 months
Correlation of EGFR, HER2, estrogen receptor and progesterone receptor immunohistochemical status as based on tumor biopsies or excisions obtained prior to this trial with objective tumor responses | up to 28 months